CLINICAL TRIAL: NCT03474952
Title: Effects of Remote Ischemic Preconditioning During Free Flap Reconstruction in Head and Neck Cancer Patients: a Randomized Controlled Trial
Brief Title: Effects of Remote Ischemic Preconditioning During Free Flap Reconstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Youn Joung Cho, MD, Clinical assistant professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RIPC during free flap
Record Dates: First submitted 2018-03-14; First posted 2018-03-23 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Remote Ischemic Preconditioning
Keywords: remote ischemic preconditioning; free flap reconstruction; tissue oxygen saturation

STUDY DESIGN:
Intervention Model Description: RIPC group and control (sham-RIPC) group
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remote ischemic preconditioning (RIPC) (Experimental): Intervention is remote ischemic preconditioning (RIPC) consists of 4 cycles of 5-min ischemia (using pneumatic cuff pressure of 200 mmHg) and subsequent 5-min reperfusion applied to upper arm.
  Interventions: Procedure: remote ischemic preconditioning (RIPC)
- Control (Sham-RIPC) (Sham Comparator): Intervention is Sham-RIPC (ischemia pressure < 10 mmHg) applied to upper arm.
  Interventions: Procedure: sham-RIPC

INTERVENTIONS:
Procedure: remote ischemic preconditioning (RIPC) — remote ischemic preconditioning consists of 4 cycles of 5-min ischemia and subsequent 5-min reperfusion using pneumatic cuff applied to upper arm
  Arms: Remote ischemic preconditioning (RIPC)
Procedure: sham-RIPC — ischemia pressure less than 10 mmHg (sham-RIPC)
  Arms: Control (Sham-RIPC)

SUMMARY:
Remote ischemic preconditioning (RIPC) has been revealed organ-protective effect in many previous clinical settings including coronary intervention or cardiovascular surgery. However its protective role during free flap reconstructive surgery in head and neck cancer patients has not yet been elucidated. The purpose of the current study is to evaluate the effect of RIPC on tissue oxygen saturation and skin temperature of the flap, as well as its organ-protective effect using Langendorff isolated heart ischemia-reperfusion model.

DETAILED DESCRIPTION:
Patients undergoing free flap reconstructive surgery for head and neck cancer will be randomized to either remote ischemic preconditioning (RIPC) group or control group. On the day of surgery, after induction of anesthesia, RIPC, consisting of 4 cycles of 5-min ischemia (using pneumatic cuff pressure of 200 mmHg) followed by 5-min reperfusion at upper arm, or sham-RIPC (pressure < 10 mmHg) will be induced in the RIPC or control group, respectively. Before completion of surgery, RIPC or sham-RIPC will be repeated. Tissue oxygen saturation and skin temperature of the flap will be recorded until postoperative day 1.

As a sub-study, blood samples will be obtained before and after RIPC/sham-RIPC. From them, plasma dialysate will be prepared to use for Langendorff isolated heart model. Myocardial infarct size of Langendorff rat heart will be compared between the groups to evaluate organ protective effect of RIPC during free flap reconstuctive surgery.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing free flap reconstructive surgery

Exclusion Criteria:

* BMI < 18, > 35 kg/m^2
* AV fistula at arm, any reason to protect arm
* vascular abnormality or discomfort at arm
* peripheral vascular disease, peripheral neuropathy, or coagulopathy
* uncontrolled diabetes mellitus
* preoperative use of beta-blocker
* history of radiation therapy
* refuse to enrol

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-04-13 (Actual); Primary Completion 2019-12-09 (Actual); Study Completion 2019-12-09 (Actual)

PRIMARY OUTCOMES:
tissue oxygen saturation | postoperative day 1
  tissue oxygen saturation of free flap

CONTACTS AND LOCATIONS:
Overall Officials: Youn Joung Cho, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Min SH, Choe SH, Kim WS, Ahn SH, Cho YJ. Effects of ischemic conditioning on head and neck free flap oxygenation: a randomized controlled trial. Sci Rep. 2022 May 17;12(1):8130. doi: 10.1038/s41598-022-12374-3. PMID 35581399